CLINICAL TRIAL: NCT03079011
Title: Randomized, Open Label, Multicentric Phase III Trial to Evaluate the Safety and Efficacy of Palbociclib in Combination With HT Driven by ctDNA ESR1 Mutation Monitoring in ER+, HER2-negative Metastatic Breast Cancer Patients
Brief Title: PAlbociclib and Circulating Tumor DNA for ESR1 Mutation Detection
Acronym: PADA-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UC-0140/1615 - UCBG3-05; 2016-004360-18 (EudraCT Number)
Record Dates: First submitted 2017-02-09; First posted 2017-03-14 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Breast Cancer
Keywords: ESR1 mutation detection, ctDNA
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Aromatase Inhibitors; Letrozole; Anastrozole; exemestane

STUDY DESIGN:
Intervention Model Description: Step 1: 1000 patients screened for circulating blood ESR1 mutation detection at regular intervals will be treated with palbociclib 125 mg once daily for 21 days followed by 7 days off (28-day cycle) + AI (letrozole, anastrozole or exemestane) administered once daily in a continuous scheme until tumor progression (assessed by RECIST) or ESR1 mutation detection
  Step 2: Up to 200 Patients with a rising circulating ESR1 mutation and without tumor progression will be randomized (1:1):
  * ARM A: no change in therapy until tumor progression (RECIST) or possibility of a cross-over (step 3)
  * ARM B: palbociclib 125 mg + fulvestrant 500 mg administered intramuscularly on D1,15 and 29 and once monthly thereafter until tumor progression (RECIST)
  * Step 3 (cross over): up to 80 patients who have been randomized in arm A will be offered to be treated by fulvestrant + palbociclib, after having progressed under AI + palbociclib until tumor progression (RECIST) under fulvestrant + palbociclib.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A- palbociclib + AI (Experimental): After randomization, the patient will be treated with palbociclib 125 mg once daily for 21 days followed by 7 days off to complete a 28-day cycle in combination with an aromatase inhibitor (letrozole, anastrozole or exemestane, according to physician's choice and according their respective summary product characteristics) administered once daily in a continuous scheme.
  Interventions: Drug: Palbociclib 125mg; Drug: Aromatase Inhibitors
- B- Palbociclib + fulvestrant (Experimental): After randomization, the patient will be treated with palbociclib 125 mg once daily for 21 days followed by 7 days off to complete a 28-day cycle in combination with fulvestrant, a selective estrogen receptor down-regulator, 500 mg administered intramuscularly on Days 1, 15, and 29 and once monthly thereafter.
  Interventions: Drug: Palbociclib 125mg; Drug: Fulvestrant Injectable Product
- Selection - Palbociclib + AI (Experimental): All patients included into the study will be treated with palbociclib 125 mg once daily for 21 days followed by 7 days off to complete a 28-day cycle in combination with an aromatase inhibitor (letrozole, anastrozole or exemestane, according to physician's choice and according their respective summary product characteristics) administered once daily in a continuous scheme
  Interventions: Drug: Palbociclib 125mg; Drug: Aromatase Inhibitors

INTERVENTIONS:
Drug: Palbociclib 125mg — Palbociclib 125 mg once daily for 21 days followed by 7 days off to complete a 28-day cycle
Drug: Aromatase Inhibitors — Letrozole: 2.5 mg once daily on a continuous scheme (tablets, per os) Anastrozole:1 mg once daily on a continuous scheme (tablets , per os) Exemestane: 25 mg once daily on a continuous scheme (tablets, per os)
  Other Names: Letrozole, Anastrozole or exemestane
  Arms: A- palbociclib + AI; Selection - Palbociclib + AI
Drug: Fulvestrant Injectable Product — 500 mg by intramuscular injection on days 1 and 15 of cycle one and then on day one of each subsequent cycle (28 days)
  Arms: B- Palbociclib + fulvestrant

SUMMARY:
This study is a randomized, open-label, multicentric, phase III trial conducted in patients receiving aromatase inhibitor and palbociclib as first line therapy for estrogen receptor (ER)-positive HER2-negative metastatic breast cancer and which aims to evaluate, at the onset of ESR1 mutations in circulating tumor DNA, the efficacy of a change of the hormone therapy (aromatase inhibitor (AI) changed to fulvestrant) combined to palbociclib, together with the safety of hormone therapy and palbociclib combination in the overall population.

ELIGIBILITY:
Inclusion Criteria:

1. Women with proven loco-regionally recurrent or metastatic adenocarcinoma of the breast not amenable to curative therapy with disease considered potentially sensitive to aromatase inhibitors Note: patients relapsing while on adjuvant tamoxifen or other non-aromatase inhibitor adjuvant endocrine therapy and patients relapsing more than one year after the end of aromatase inhibitor adjuvant therapy are eligible for the present study;
2. Age ≥18 years;
3. Life expectancy >3 months;
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2;
5. Estrogen Receptor (ER)-positive and HER2-negative breast cancer. Where available, assessment of Estrogen Receptor status should be based on the most recent tumor sample; to be considered as ER-positive, the most recent breast cancer tissue examined must display at least 10% of cancer cells with positive ER staining;
6. Tumor block (primary tumor or metastasis) available;
7. No prior systemic anti-cancer therapy for metastatic or advanced disease (chemotherapy, targeted therapy or hormone therapy); prior initiation of LHRH agonist or bone-directed agents is however allowed);
8. Menopausal patients or patients with suppressed ovarian function

   * Women with bilateral oophorectomy
   * Postmenopausal women, as defined by any of the following criteria:

     * Age 60 or over;
     * Age 50 to 59 years and meets one of the following criteria:

       * Amenorrhea for ≥24 months and follicle-stimulating hormone within the postmenopausal range;
       * patients with hysterectomy or chemotherapy-induced amenorrhea must display follicle-stimulating hormone within the postmenopausal range;
   * Other women, provided they are being treated with monthly LHRH analogues (first injection performed ≥7 days before the treatment initiation) and are willing to continue to receive LHRH agonist therapy for the duration of the trial;
9. Patients may have measurable (according to Response Evaluation Criterion in Solid Tumors (RECIST v1.1) or not measurable disease

   * Patients with only blastic bone lesions are not eligible;
   * Patients with only pleural, cardiac or peritoneal effusion or meningeal carcinomatosis are not eligible;
10. Adequate organ and marrow function as defined below:

    * Hemoglobin ≥90 g/L
    * Absolute neutrophil count ≥1.5 g/L
    * Platelet count ≥100 g/L
    * Serum bilirubin ≤1.5 × upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome.
    * ALT and AST ≤3 × ULN;
    * Alkaline phosphatase ≤2.5 x ULN (≤5.0 x ULN if bone or liver metastases present)
    * Serum creatinine ≤1.5 × ULN or calculated creatinine clearance ≥ 60 mL/min as determined by Cockcroft-Gault (using actual body weight) formula for females [creatinine clearance =Weight (kg) × (140 - Age) × 0.85 (mL/min)/ (72 × serum creatinine (mg/dL))
11. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and any protocol-related procedures including screening evaluations;
12. Resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to NCI CTCAE version 4.03 Grade 1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion);
13. Written informed consent obtained prior to performing any protocol-related procedures including screening evaluations;
14. Patient affiliated to a social security system.

Exclusion Criteria:

1. Locally advanced breast cancer or loco-regional relapse amenable for any treatment with curative intent;
2. Her2-positive or equivocal tumor status either on the primary or on the recurrent tumor, defined as IHC3+, Fish/Cish amplified or Fish/Cish equivocal according to the ASCO2015 criteria;
3. Prior endocrine therapy in the metastatic setting is not allowed;
4. Prior treatment with any CDK 4/6 inhibitor in the adjuvant or metastatic setting (neoadjuvant/preoperative treatment is allowed); however, prior therapy with another targeted treatment in the adjuvant setting is allowed;
5. Visceral crisis: Advanced, symptomatic, visceral spread that is at risk of life-threatening complication in the short term and that requires chemotherapy;
6. Any major surgery (defined as requiring general anaesthesia) or significant traumatic injury within 4 weeks of treatment initiation or patients that may require major surgery during the course of the study; however, surgical diagnostic procedure is allowed (even if performed under general anaesthesia);
7. Known, active bleeding diathesis;
8. Any serious known concomitant systemic disorder (e.g. known active infection including HIV, or cardiac disease) incompatible with the study (at the discretion of investigator), previous history of bleeding diathesis, or anti-coagulation treatment (the use of low molecular weight heparin is allowed);
9. Patients unable to swallow tablets;
10. History of mal-absorption syndrome or other condition that would interfere with enteral absorption;
11. Chronic daily treatment with corticosteroids with a dose of ≥10 mg/day methylprednisolone equivalent (excluding inhaled steroids);
12. Known active uncontrolled or symptomatic central nervous system (CNS) metastases, carcinomatous meningitis, or leptomeningeal disease as indicated by clinical symptoms, cerebral oedema, and/or progressive growth. Patients with a history of CNS metastases or cord compression are eligible if they have been definitively treated with local therapy (e.g., radiotherapy, stereotactic surgery) and are clinically stable and off anticonvulsants and steroids for at least 4 weeks before treatment start;
13. Known hypersensitivity to letrozole, anastrozole, exemestane, fulvestrant, palbociclib or any of their excipients;
14. Uncontrolled electrolyte disorders that can compound the effects of a QTc prolonging drug (e.g., hypocalcemia, hypokalemia, hypomagnesemia);
15. Patients treated within the last 7 days prior to treatment start in the trial with drug that are known to be CYP3A4 inhibitors, drugs that are known to be CIP3A4 inducers, who underwent a grapefruit cure;
16. Patients already included in another therapeutic trial evaluating an investigational medicinal product or having received an investigational medicinal product within 3 months;
17. History of previous:

    * Any other stage II, III, IV cancer within 5 years preceding patient enrollment in the trial - however, multiple primary breast cancers (controlateral/ipsilateral cancers/local relapses) are allowed pending all tumor masses were ER+;
    * Any history of hematological malignancy;
18. Persons deprived of their freedom or under guardianship or incapable of giving consent;
19. Pregnancy or lactation period. Women of childbearing potential must implement adequate non-hormonal contraceptive measures (barrier methods, intrauterine contraceptive devices, sterilization; LHRH agonist cannot be considered as an efficient contraceptive measure) during study treatment and for 90 days after discontinuation. A serum pregnancy test must be negative in premenopausal women or women with amenorrhea of less than 12 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1017 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent Adverse Events | Throughout study completion, up to 4 years
  Global safety of the combination of palbociclib + endocrine therapy in the whole population, with focus on hematological toxicities.
  Safety will be assessed by the collection of grade ≥3 adverse events, using the Common Terminology Criteria for Adverse Events (CTCAE), version 4.03 - in all included patients.
Progression-free survival (Step 2) | From randomization to disease progression or death, up to 4 years
  To assess whether a change of the hormone therapy associated with palbociclib will benefit patients for whom rising ESR1 mutations are detected during treatment with palbociclib and aromatase inhibitor.
  Progression-Free Survival (PFS) will be measured from the time of randomization to the time of tumor progression (as assessed by the investigator per RECIST v1.1) or death (whichever comes first) - in randomized patients.

SECONDARY OUTCOMES:
Progression-free survival (step 3) | From cross-over, up to 4 years
  To assess PFS in patients undergoing a cross-over following RECIST tumor progression in Arm A, from the start of crossover.
  Progression-Free Survival will be measured from the time of cross-over to the time of tumor progression (as assessed by the investigator per RECIST 1.1) or death (whichever comes first) - in all patients with crossover
Progression-free survival (step 1&2) | From inclusion, up to 4 years
  To report efficacy (PFS based on RECIST) of palbociclib combined with hormone therapy (aromatase inhibitor or fulvestrant), from the date of initial inclusion into the trial.
  Progression-Free Survival will be measured from the time of inclusion to the time of tumor progression (as assessed by the investigator per RECIST 1.1) or death (whichever comes first) - in all included patients including those who switched to fulvestrant.
Time to strategy failure from randomization (Step 2 and 3) | From randomization, up to 4 years
  To assess whether the early switch (switch following ESR1 mutations increase) to fulvestrant contributes to a longer time to strategy failure than a late switch (cross-over following RECIST tumor progression).
  Time to strategy failure will be measured from the time of randomization until palbociclib+endocrine therapy discontinuation or death (whichever comes first) - in all randomized patients.
Chemotherapy-free survival (Step 2 and 3) | From randomization, up to 4 years
  To assess whether the early switch (following ESR1 mutations increase) to fulvestrant contributes a longer chemotherapy-free survival than a late switch (cross-over following RECIST tumor progression).
  Chemotherapy-free survival will be measured from the time of randomization until the date of chemotherapy initiation or death (whichever comes first) - in all randomized patients.
Incidence of treatment-emergent extra-hematological Adverse Events | Throughout study completion, up to 4 years
  To obtain additional safety data in a broad patient population treated with palbociclib and hormone therapy (aromatase inhibitor or fulvestrant) in a general Description of all extra-hematological grade ≥3 toxicities and SAEs incidence rate in the overall population and each treatment step
Quality of life by quality of life questionnaire (QLQ)-C30 | From inclusion and every 2 months until disease progression, up to 2 years
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Other line of therapy | Throughout study completion, up to 4 years
  To report the anti-cancer treatments received after the first line therapy.
Overall Survival | Throughout study completion, up to 4 years
  The overall survival is the length of time from inclusion that patients enrolled in the study are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: François-Clément BIDARD, MD PhD, Principal Investigator — Institut Curie; Suzette DELALOGE, MD PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris; Anne-Claire HARDY BESSARD, MD, Principal Investigator — Centre Armoricain d'Oncologie
Locations (82):
- France (82):
  - Centre Hospitalier Universitaire, Amiens
  - Clinique de l'Europe, Amiens
  - Institut de Cancérologie de l'Ouest - Site Paul Papin, Angers
  - Centre Hospitalier d'Auxerre, Auxerre
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier de Beauvais, Beauvais
  - Centre Hospitalier de Blois, Blois
  - Clinique Tivoli Ducos, Bordeaux
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre Hospitalier de boulogne sur Mer, Boulogne-sur-Mer
  - Centre Hospitalier Fleyriat, Bourg-en-Bresse
  - CHRU Morvan, Brest
  - Clinique PASTEUR-CFRO, Brest
  - Centre Francois Baclesse, Caen
  - Centre Hospitalier René Dubos, Cergy-Pontoise
  - Medipole de Savoie, Challes-les-Eaux
  - Centre Hôpital Sainte Marie, Chalon-sur-Saône
  - CH William Morey, Chalon-sur-Saône
  - Centre Hospitalier Métropole de Savoie, Chambéry
  - Centre Hospitalier de Cholet, Cholet
  - Centre Jean Perrin, Clermont-Ferrand
  - Pôle Santé République, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - CHI Fréjus St-Raphaël, Fréjus
  - Institut Daniel Hollard - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Centre Hospitalier Départemental de Vendée, La Roche-sur-Yon
  - Clinique du Cap d'Or, La Seyne-sur-Mer
  - Centre Hospitalier de Versailles, Le Chesnay
  - Centre Hospitalier le Mans, Le Mans
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - CHU Dupuytren, Limoges
  - Clinique François Chénieux, Limoges
  - Centre Hospitalier Bretagne Sud, Lorient
  - Centre Leon Berard, Lyon
  - Clinique de la Sauvegarde, Lyon
  - Hôpital privé Jean Mermoz, Lyon
  - Hôpital Européen Marseille, Marseille
  - Hôpital Saint Joseph, Marseille
  - Institut Paoli Calmettes, Marseille
  - Centre d'Oncologie radiothérapie de Macon, Mâcon
  - Clinique Claude Bernard, Metz
  - Centre Hospitalier ANNECY GENEVOIS, Metz-Tessy
  - CH Mont de Marsan, Mont-de-Marsan
  - Centre Hospitalier Montceau les mines, Montceau-les-Mines
  - ICM - Val d'Aurelle, Montpellier
  - Centre d'Oncologie de Gentilly, Nancy
  - Hopital Privé du Confluent, Nantes
  - Centre Antoine Lacassagne, Nice
  - Centre ONCOGARD - Institut de Cancérologie du Gard, Nîmes
  - Institut Curie, Paris
  - Hopital Diaconesses-Croix Saint Simon, Paris
  - Hopital Européen Georges Pompidou, Paris
  - Saint Louis Hospital, Paris
  - Centre Hospitalier de Pau, Pau
  - Centre Catalan d'Oncologie, Perpignan
  - Polyclinique Francheville, Périgueux
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CARIO - Centre Armoricain Radiothérapie Imagerie Médicale et Oncologi, Plérin
  - Centre Hospitalier de Cornouaille, Quimper
  - Clinique de la Croix du Sud, Quint-Fonsegrives
  - Centre Eugène Marquis, Rennes
  - Centre de radiothérapie et d'oncologie médicale LE-CROME, Ris-Orangis
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier Saint-Brieuc, Saint-Brieuc
  - Institut Curie - Hôpital René Huguenin, Saint-Cloud
  - CHP Saint Grégoire, Saint-Grégoire
  - Institut de Cancérologie de l'Ouest - Site René Gauducheau, Saint-Herblain
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - Institut de cancérologie lucien Neuwith, Saint-Priest-en-Jarez
  - Centre Hospitalier de Broussais, St-Malo
  - Centre Paul Stauss, Strasbourg
  - Clinique de l'Orangerie, Strasbourg
  - Clinique Sainte Anne, Strasbourg
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Hôpitaux du Léman, Thonon-les-Bains
  - Clinique Pasteur, Toulouse
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier de Tours - Hopital Bretonneau, Tours
  - Centre Hospitalier Bretagne Atlantique, Vannes
  - UNEOS Site Hôpital Robert Schuman, Vantoux
  - Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Bidard FC, Hardy-Bessard AC, Dalenc F, Bachelot T, Pierga JY, de la Motte Rouge T, Sabatier R, Dubot C, Frenel JS, Ferrero JM, Ladoire S, Levy C, Mouret-Reynier MA, Lortholary A, Grenier J, Chakiba C, Stefani L, Plaza JE, Clatot F, Teixeira L, D'Hondt V, Vegas H, Derbel O, Garnier-Tixidre C, Canon JL, Pistilli B, Andre F, Arnould L, Pradines A, Bieche I, Callens C, Lemonnier J, Berger F, Delaloge S; PADA-1 investigators. Switch to fulvestrant and palbociclib versus no switch in advanced breast cancer with rising ESR1 mutation during aromatase inhibitor and palbociclib therapy (PADA-1): a randomised, open-label, multicentre, phase 3 trial. Lancet Oncol. 2022 Nov;23(11):1367-1377. doi: 10.1016/S1470-2045(22)00555-1. Epub 2022 Sep 29. PMID 36183733
- [Derived] Berger F, Marce M, Delaloge S, Hardy-Bessard AC, Bachelot T, Bieche I, Pradines A, De La Motte Rouge T, Canon JL, Andre F, Arnould L, Clatot F, Lemonnier J, Marques S, Bidard FC; PADA-1 investigators. Randomised, open-label, multicentric phase III trial to evaluate the safety and efficacy of palbociclib in combination with endocrine therapy, guided by ESR1 mutation monitoring in oestrogen receptor-positive, HER2-negative metastatic breast cancer patients: study design of PADA-1. BMJ Open. 2022 Mar 3;12(3):e055821. doi: 10.1136/bmjopen-2021-055821. PMID 35241469